CLINICAL TRIAL: NCT00172471
Title: The Relationship Between Sleep Disorders and Cytokine Levels Among Hemodialysis and Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700775
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2004-12

CONDITIONS: Renal Failure; Sleep Disorder; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Sleep disorders are common in patients with end-stage renal disease on both hemodialysis and peritoneal dialysis and are associated with significant medical, psychological and social disturbances. Numerous factors have been suggested as contributing to or associated with the high prevalence of sleep disturbance in this population.

Increasing evidence suggests that cytokines are involved in the regulation of sleep and wakefulness and that the communication between the sleep and the immune system is bi-directional. Blood-dialyzer or peritoneum-dialysate interaction during dialysis therapy has the potential to activate mononuclear cells leading to production of inflammatory cytokines. These cytokines are believed to play a significant role in dialysis-associated morbidity and mortality. Nevertheless, a cytokine overproduction may alter sleep pattern in chronic dialyzed patients, thus explaining the presence of sleep disorders in these patients. In the other way, sleep loss may have effects on immune process and secretion of cytokines in chronic dialyzed patients. The purpose of this study was to examine the relationship between quality of sleep and serum cytokine levels in hemodialysis and peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* ESRD Patients with hemodialysis or peritoneal dialysis

Exclusion Criteria:

* Malignancy, hospitalization, infection, inflammation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jenq-Wen Huang, MD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Division of Nephrology, Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan